CLINICAL TRIAL: NCT06559098
Title: Vibrotactile Coordinated Reset (vCR) for the Treatment of Advanced Parkinson's Disease Patients Who Have Previously Received vCR Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vivek P. Buch, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71579
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinsons; vibrotactile stimulation; vibration; PD; Non-invasive
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Patients who have previously received non invasive vibrotactile stimulation meant to reduce symptoms of Parkinson's disease will be enrolled and will be asked to stimulate with the Stanford Coordinated Reset (CR) glove
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stimulation (Experimental): Patients who were previously enrolled in a vibrotactile study meant to reduce symptoms associated with Parkinson's disease will be enrolled in the study and will be asked to stimulate with the Stanford Coordinated Reset(CR) glove in sessions that last 2 hours. Sessions may be daily or a few times weekly depending on the needs of the patient.
  Interventions: Device: Vibrotactile coordinated reset (vCR)

INTERVENTIONS:
Device: Vibrotactile coordinated reset (vCR) — Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. A specific pattern of vibration to each fingertip is delivered which theoretically disrupts abnormal synchrony in the brain
  Other Names: Stanford Coordinated Reset Glove

SUMMARY:
The purpose of this study is to test the efficacy of vibrotactile coordinated reset(vCR) stimulation on human subject participants with advanced stage Parkinson's Disease who have previously received vCR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any adult age 18 and older
* Idiopathic Parkinson's Symptoms between Hoehn and Yahr stages 2 to 4
* Fluent in English
* If patient is on medication that affects brain function or alters Electroencephalography (EEG) activity, the patient must feel comfortable going off this medication prior to EEG recording
* Appropriate social support if required during an off state.
* Comfortable with technology; can use a computer, check email, and access the internet; can initiate and engage in a virtual meeting for training and monitoring purposes.
* Feels comfortable going off Parkinson's Disease(PD) related medication during in person study visits
* Lives in the United States
* Having previously been enrolled in a vCR pilot study

Exclusion Criteria:

* Any significant neuro-psychiatric problems, including acute confusional state, ongoing psychosis, or suicidal tendencies
* Any current drug or alcohol abuse.
* Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
* Pregnancy, breast-feeding or wanting to become pregnant
* Physical limitations unrelated to PD that would affect motor ratings
* Craniotomy
* Brain surgery
* Patient is unable to communicate properly with staff (i.e., severe speech problems)
* Excessive drooling
* A type of hairstyle that would impede the use of an EEG cap
* Sensory abnormalities of the fingertips
* Patient is taking a medication that may cause significant withdrawal effects.
* Presence or diagnosis of Essential Tremor, psychogenetic tremor, functional tremor and any other non- pathological or non-Parkinsonian tremors

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS III) off medication | Baseline, 3Months,6 Months, 9 Months 12 Months, 18 Months, 24 Months
  This scale measures motor ability within Parkinson's patients. For part 3, the scales minimum values is 0 and max value is 132. Higher scores indicate more impaired motor ability, while lower scores indicate less impaired motor ability. A score of 0 indicates no motor impairment.

SECONDARY OUTCOMES:
Levodopa equivalent daily dose (LEDD) daily change from baseline to 24 months | 24 months
  LEDD is calculated as a daily sum of levodopa in each Parkinson's medication
Parkinson's disease quality of life questionnaire-39 (PDQ-39) | 24 months
  The PD Quality of Life Questionnaire-39 (PDQ-39) is a self-report questionnaire that examines health related difficulties specific to PD in eight quality of life categories within the last month. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100, with higher % indicating more health problems.
Freezing of Gait Questionnaire (FOG) change | 24 months
  The Freezing of Gait questionnaire (FOG) assesses severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning). The FOG is comprised of 6 questions measured on a 0 to 4 scale (where 0 is normal and 4 represents severe abnormalities). The scores are summed together with 0 representing the best possible score and 24 representing the worst possible score.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 1 change | 24 months
  The MDS-UPDRS part 1 focuses on non-motor symptoms, such as dementia, depression, and psychosis. The total summed score ranges from 0-52 with higher scores indicating increased non-motor impairment.
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 2 | 24 months
  The MDS-UPDRS part 2 focuses on the patient's ability to perform daily motor activities including dressing, grooming, and using utensils. The total summed score ranges from 0-52 with higher scores indicating increased daily motor impairment
Movement disorders unified Parkinson's rating scale (MDS-UPDRS) part 4 change | 24 months
  The MDS-UPDRS 4 focuses on Measures the complications of treatment, e.g. dyskinesias and motor fluctuations. The total summed score ranges from 0-24 with higher scores indicating increased motor complications.
Communicative Participation Item Bank (CPIB; Short Form) | 24 months
  The CPIB is a questionnaire that measures speech complications. The questionnaire is scored from 0 to 30, with a higher score indicating increased speech difficulties.
Voice Handicap Index (VHI-10) | 24 months
  This questionnaire can be filled out by patients and assesses the impact that voice problems and limitations have on the individual's overall daily function. Questionnaire is scored from 0 to 40, with a higher score indicating increased speech difficulties.
Spontaneous Electroencephalography beta band power change | 24 months
  Patients will be recorded while receiving vibrotactile stimulation. The Beta Band (13-30Hz) power spectral density (PSD) will be of interest. The units of the power spectral density are micro-Volts-squared per Hz. Increases in Beta band PSD are associated with motor impairment in Parkinson's disease, while decreases in the beta band are associated with motor improvement.
Parkinson's disease cognitive functional rating scale (PD-CFRS) | 24 months
  The PD-CFRS capture subjective daily functional cognitive decline among patients with Parkinson's disease over the past 2 weeks. The scale ranges from 0 to 24, with higher scores indicative of cognitive decline.
Device calibration | 24 months
  Participants will be assessed for their perceptive threshold of vibration, or the lowest vibration amplitude perceived. This is determined by adjusting the amplitude of the experimental device.